CLINICAL TRIAL: NCT01453478
Title: A Single Centre, 5-Period, Randomized Study To Evaluate The Relative Bioavailability Of An Immediate Release Tablet Formulation And Prototype Bioenhanced Formulations Of GSK1325756 In Healthy Elderly Subjects During Suppression Of Gastric Acid Secretion
Brief Title: A Study to Look at How GSK1325756 is Taken up by the Body When Given by Mouth When Stomach Acid is Reduced
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 115550
Record Dates: First submitted 2011-10-13; First posted 2011-10-18 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — danirixin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- GSK1325756 Immediate Release 50 mg (Experimental): Administered to volunteers in the fasted and fed states
  Interventions: Drug: GSK1325756
- GSK1325756 Bioenhanced Formulation 1 50 mg (Experimental): Administered to volunteers in the fasted and/or fed states
  Interventions: Drug: GSK1325756
- GSK1325756 Bioenhanced Formulation 2 50 mg (Experimental): Administered to volunteers in the fasted and/or fed states
  Interventions: Drug: GSK1325756

INTERVENTIONS:
Drug: GSK1325756 — CXCR2 antagonist

SUMMARY:
This is a Phase I study to assess the combined effects of food and suppression of gastric acid secretion on the relative bioavailability of an immediate release (IR) tablet formulation and prototype bioenhanced formulations of GSK1325756, an oral interleukin 8 receptor (IL8R also known as CXCR2) antagonist. The objectives are to understand if the co-administration of food enhances absorption and the inter-subject variability for the current GSK1325756 IR tablet under fed state proton pump inhibitor (PPI) conditions and secondly to assess whether two proposed bioenhanced formulations offer any improvement over the current GSK1325756 IR formulation under PPI conditions.

This open-label, randomized, 5-period crossover study will be completed in a single cohort of subjects, with an interim analysis after completion of Treatment Period 4. During Treatment Periods 1 to 4, subjects will be randomized to receive GSK1325756 50 mg IR in the fed state, GSK1325756 50 mg IR in the fasted state, GSK1325756 Bioenhanced Formulation 1 in the fasted state, and GSK1325756 Bioenhanced Formulation 2 in the fasted state. Progression to Treatment Period 5 and the choice of bioenhanced formulation for dosing in this treatment period will be dependent on the findings of an interim analysis of the pharmacokinetic profile and relative bioavailability of each formulation following completion of Treatment Periods 1 to 4. In Treatment Period 5, subjects will receive the selected GSK1325756 bioenhanced formulation in the fed state.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the relative bioavailability, including the inter-subject variability, of the immediate release (IR) tablet used for the previous Phase I studies and 2 prototype bioenhanced tablet formulations of GSK1325756 in healthy elderly male and female subjects under fed and fasted states during suppression of gastric acid secretion (concomitant omeprazole, 20 mg, once daily (QD)). Secondary objectives include provision of information on the oral pharmacokinetic (PK) of GSK1325756 in the elderly under different dosing conditions during suppression of gastric acid secretion, and additional safety and tolerability information for oral administration of GSK1325756 in elderly subjects.

The current study will provide an understanding of the PK of three formulations of GSK1325756 during gastric acid suppression in a population of 65 to 80 year old healthy adult subjects. The effect of food on the PK of each GSK1325756 formulation will also be addressed in this population. The outcome of this study is likely to guide selection of the most appropriate formulation/dosing regimen for future studies.

The completed clinical studies demonstrated that to minimize inter-subject variability of the exposure to GSK1325756, the current formulation needs to be administered with food, particularly in elderly subjects. This does not preclude development of the current formulation, but is not ideal, particularly if twice daily administration is needed in chronic obstructive pulmonary disease (COPD) patients and for elderly subjects in which food intake can be variable. In addition, the inter-subject variability in exposure with the current formulation when given with omeprazole in the fasted state is not acceptable. This is likely due to the need for a low pH (acid level) (pH < 2) gastric environment, particularly in the fasted state, to allow for sufficient solubilization of the GSK1325756 prior to transport to the small intestine where it is absorbed. Thus, this study is being conducted for the following reasons: (1) to determine if the current formulation results in acceptable exposure and inter-subject variability if given with food in subjects in which gastric acid secretion is suppressed with omeprazole and (2) to determine if a bio-enhanced formulation can provide an acceptable exposure profile and acceptable inter-subject variability in the fasted state in subjects in which gastric acid is suppressed. This information will be important in helping to determine the appropriate formulation and dosing regimen for progression to studies in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-childbearing potential female who, at the time of signing the informed consent, are aged between 65 and 80 years (inclusive). Non-childbearing potential is defined as pre-menopausal females with a documented tubal ligation or hysterectomy or postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] greater than 40 milli-international units per milliliter MlU/mL) and estradiol less than 40 picograms per milliliter (pg/mL) [less than 147 picomoles per liter (pmol/L)] is confirmatory).
* Healthy, as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the investigator and the GlaxoSmithKline (GSK) Medical Monitor agree that the finding is unlikely to introduce risk factors and will not interfere with the study procedures and objectives.
* Aspartate aminotransferase (AST), alanine transaminase (ALT), alkaline phosphatase and bilirubin less than or equal to 1.5 times the upper limit of normal (ULN) (isolated bilirubin greater than 1.5 times the ULN is acceptable if bilirubin is fractionated and direct bilirubin is less than 35 percent (%)).
* Resting blood pressure of less than or equal to 160/95 millimeters of mercury (mm Hg), irrespective of anti-hypertensive medication status for the subject.
* Body weight greater than or equal to 60 kilograms (kg) for men and greater than or equal to 45 kg for women; body mass index within the range 19 to 32 kiligrams per meter squared (kg/m2) (inclusive).
* Male subjects with female partners of child-bearing potential must agree to use two of the following acceptable forms of contraception methods, one of which must be a barrier method, from screening until 12 weeks after the last dose of study treatment: 1) Established use of oral, injected or implanted methods of contraception. (The decision to allow use of hormonal contraceptives should be based on the investigational medicinal product's metabolism and potential for interactions, pharmacology and adverse event profile e.g., vomiting) 2) Placement of an intrauterine device or system 3) Barrier method such as a condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository. Barrier contraceptives must always be supplemented with the use of a spermicide, which are not a barrier method and therefore should not be used alone 4) Male sterilization 5) True abstinence is acceptable when in line with the preferred and usual lifestyle of the subject. If a subject is not usually sexually active but becomes active, they should, with their partner, use two of the contraceptive methods listed above.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study Hepatitis B surface antigen (HBsAg) or positive Hepatitis C antibody (HCV Ab) result within 3 months of screening.
* A positive pre-study drug/alcohol screen, with the exception of a positive result considered by the investigator to be directly attributable to prescription medication approved for subject use during the study.
* A positive test for human immunodeficiency virus (HIV) antibody.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of greater than 21 units for males or greater than 14 units for females. One unit is equivalent to 8 grams of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Positive urine beta-human chorionic gonadotropin (β-hCG) test at screening or prior to first dose for female subjects.
* Screening QT interval analysed by Bazett correction (QTcB) greater than 450 msec, PR interval outside the range 120 to 220 msec or an ECG that is not suitable for QT measurements (e.g., poorly defined termination of T wave).
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 3 months, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study treatment until completion of the post-study medical, unless in the opinion of the investigator and GlaxoSmithKline (GSK) Medical Monitor, the medication will not interfere with the study procedures or compromise subject safety; examples are anti-hypertensive medication for at least 3 months prior to the screening visit and lipid-lowering medications (statins or fibrates) for at least 3 months prior to the screening visit.
* History of sensitivity to any of the study treatments, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 milliliters (mL) within a 3-month period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* Exhaled breath carbon monoxide levels indicative of smoking (greater than 10 parts per million at screening), or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Consumption of red wine, Seville oranges, grapefruit or grapefruit juice and/or pummelos, citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study treatment until collection of the final blood sample during each treatment period.
* Galactose intolerance, Lapp-lactase deficiency or glucose-galactose malabsorption.
* Direct involvement in the conduct of the study, or relative of any person directly involved in the conduct of the study.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-10-12 (Actual); Primary Completion 2011-12-19 (Actual); Study Completion 2011-12-19 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | Forty eight hour period following dose
  For determination of Area Under the blood concentration time Curve (AUC) for GSK1325756

SECONDARY OUTCOMES:
Pharmacokinetics | Forty eight hour period following dose
  For determination of GSK1325756 pharmacokinetic parameters other than Area Under the blood concentration time Curve (AUC)
Safety and tolerability information | Study Duration
  Adverse event (AE) reporting, vital signs, electrocardiograms (ECGs), changes in clinical laboratory parameters, and changes in clinical signs and symptoms from physical examination, as data permit.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 115550 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115550?search=study&study_ids=115550#rs
- Available data/document: Statistical Analysis Plan: 115550 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115550 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115550 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115550 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115550 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115550 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115550 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register